CLINICAL TRIAL: NCT02702726
Title: The Oil, Fats and Oleogel (OFO) Study: Effects of Dietary Fats, Ingested in Two Physical Forms, on Acute Human Energy Balance, Appetitive and Glycemic Responses
Brief Title: The Oil, Fats and Oleogel Study
Acronym: OFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015/01093
Record Dates: First submitted 2016-02-29; First posted 2016-03-09 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Glycaemic Response and Energy Balance
MeSH Terms: interventions — Coconut Oil; Sunflower Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Congee and juice only (No Intervention): Control breakfast providing 50g carbohydrate
- Congee and juice with coconut gel (Active Comparator): Control breakfast, plus 25g coconut oleogel (solid)
  Interventions: Other: Congee and juice with coconut gel
- Congee and juice with coconut oil (Active Comparator): Control breakfast, plus 25g coconut oil (liquid)
  Interventions: Other: Congee and juice with coconut oil
- Congee and juice with sunflower gel (Active Comparator): Control breakfast, plus 25g sunflower oleogel (solid)
  Interventions: Other: Congee and juice with sunflower gel
- Congee and juice with sunflower oil (Active Comparator): Control breakfast, plus 25g sunflower oil (liquid)
  Interventions: Other: Congee and juice with sunflower oil

INTERVENTIONS:
Other: Congee and juice with coconut gel — 25g coconut oleogel
  Arms: Congee and juice with coconut gel
Other: Congee and juice with coconut oil — 25g coconut oil
  Arms: Congee and juice with coconut oil
Other: Congee and juice with sunflower gel — 25g sunflower oleogel
  Arms: Congee and juice with sunflower gel
Other: Congee and juice with sunflower oil — 25g sunflower oil
  Arms: Congee and juice with sunflower oil

SUMMARY:
The aim of this study is to compare the effects of dietary fats, ingested in two physical forms, on acute energy balance, appetitive, and glycemic responses of healthy normal (BMI 18-24.9 kgm-2) or overweight (BMI>25kgm-2) adults.

DETAILED DESCRIPTION:
This will be a randomised, crossover study. Randomisation will be performed with an online randomisation software (www.randomizer.org). Participants will be screened (1 screening visit) and attend five test visits conducted in a whole room calorimeter (WRC). During each test visit, participants will arrive at the laboratory after an overnight fast, enter the WRC and rest for 15 minutes in a supine position,have their resting energy expenditure (REE) measured for 30 minutes and consume congee and juice alone(control), or with one of the 4 dietary fats: sunflower oil (SO) or gel (SG) and coconut oil (CO) or gel (CG) (total 5 test visits). Post-meal energy expenditure, fat oxidation, glycemia and appetite (visual analog scales) will be measured continuously for 3 hours in WRC, followed by a meal challenge where participants will eat until sated. Participants will return and repeat the protocol until all fat types and forms are completed.

ELIGIBILITY:
Exclusion Criteria:

* People with major chronic disease such as heart disease, cancer, hypertension or diabetes mellitus
* People with known food allergies, due to potential traces of allergens found in the commercially available food product used in our study (Knorr's instant congee)
* People who are claustrophobic
* Individuals who are taking insulin or drugs known to affect glucose metabolism, appetite, and body fat distribution
* Have weight change of >5kg in the past 3 months
* People with a major medical or surgical event requiring hospitalization within the preceding three months
* People who are on a weight loss regime
* Individuals with the presence of disease or drugs which influence digestion and absorption of nutrients

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
180-min postprandial energy expenditure (kJ/min over 180 minutes and total kJ/180-min session) measured by an indirect ventilated-hood calorimeter | 180 minutes
  Gaseous exchanges obtained from the indirect calorimeter (volume of oxygen consumed and volume of carbon dioxide produced) will be used to calculate energy expenditure using the Weir equation: EE = 3.9 VO2 + 1.1 VCO2 [Weir, J. B. (1949). "New methods for calculating metabolic rate with special reference to protein metabolism." Journal of Physiology 109(1): 1-9]
180-min postprandial carbohydrate and fat oxidation (kJ/min over 180 minutes and total kJ and total grams during each session) measured by an indirect ventilated-hood calorimeter | 180 minutes
  Gaseous exchanges obtained from the indirect calorimeter (volume of oxygen consumed and volume of carbon dioxide produced) will be used to calculate energy expenditure using the Frayn equations: carbohydrate oxidation = 4.55 VCO2 - 3.21 VO2; fat oxidation = 1.67 VO2 - 1.67 VCO2 [Frayn, K. N. (1983). "Calculation of substrate oxidation rates in vivo from gaseous exchange." Journal of Applied Physiology 55(2): 628-634]
Post-test-meal capillary blood glucose (mmol/L) at 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes | 180 minutes
  Capillary blood glucose will be assessed at 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes using a Hemocue system (HemoCue Glucose 201 RT Systems, Helsingborg, Sweden)

SECONDARY OUTCOMES:
Post-test-meal subjective appetite measurements at 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes | 180 minutes
  Appetite ratings will be collected at 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes after test meal consumption using a previously validated visual analog scales [Flint, A., A. Raben, J. E. Blundell and A. Astrup (2000). "Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies." International Journal of Obesity 24(1): 38-48]
Free-living food intake after completion of test session | 180 minutes
  Participants will be asked to keep a food record that document the types and amount of food and beverage they consume after they leave the research centre, until they go to bed on the same day. Data will be analysed using nutrient analysis software.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Not applicable for this study

REFERENCES:
- [Derived] Tan SY, Peh E, Lau E, Marangoni AG, Henry CJ. Physical Form of Dietary Fat Alters Postprandial Substrate Utilization and Glycemic Response in Healthy Chinese Men. J Nutr. 2017 Jun;147(6):1138-1144. doi: 10.3945/jn.116.246728. Epub 2017 May 10. PMID 28490674